CLINICAL TRIAL: NCT05473572
Title: The Effect of Stuttering Remediation Exercises on Cortical Auditory Evoked Potentials in School Age Children Who Stutter
Brief Title: Effect of Stuttering Remediation Exercises on Cortical Auditory Evoked Potentials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alaa Mamdouh (Other)
Responsible Party: Sponsor-Investigator, Alaa Mamdouh, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0201568; 00012098 (Other: IRB); 00018699 (Other: FWA)
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Developmental Stuttering; Evoked Potentials Auditory
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Intervention Model Description: two groups group of children who stutter group of children who do not stutter
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children who stutter (Experimental): Measuring stuttering severity and cortical auditory evoked potentials in a group of children who stutter then they will receive fluency shaping exercises for a period range from 2-4 months. Reassessment of cortical auditory evoked potentials and stuttering severity after the specified period
  Interventions: Behavioral: Fluency shaping exercises
- children who do not stutter (No Intervention): Measuring cortical auditory evoked potentials as a comparison group

INTERVENTIONS:
Behavioral: Fluency shaping exercises — Training for prolonged speech, easy onset, light contact and abdominal breathing moving from the level of single words till using short sentences describing pictures
  Arms: Children who stutter

SUMMARY:
studying how the cortical auditory evoked potentials differ in children who stutter from who do not stutter and how these potentials change with therapy

DETAILED DESCRIPTION:
Measuring amplitude and latency of P1, N1, P2 N2 between a group with developmental stuttering and a control group with no stuttering at baseline. Recording the potentials through passive listening to a 60dB stimulus and active speaking, describing pictures and rapid naming.

Assigning the group with stuttering to remediation exercises using fluency shaping program for 2 to 4 months then remeasuring amplitude and latency of the previously mentioned potentials.

ELIGIBILITY:
Inclusion criteria:

* Patients with developmental stuttering
* Normal hearing and vision.
* Adequate language for age.

Exclusion criteria:

* Known history of epileptic fits.
* Intellectual disability and other neurological deficits.
* Cluttering

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Difference in latency of cortical auditory evoked potentials in children with stuttering compared to children who do do not stutter | baseline: before intervention
  Measuring latency in millisecond of P1, N1 using the commercial system (Interacoustic Eclipse TM) device during passive listening to a 60dB auditory stimulus and active speaking conditions
Change in latency of cortical auditory evoked potentials in children with stuttering due to stuttering intervention program | immediately after intervention
  Measuring latency in millisecond of P1, N1 in the group who stutter after intervention using the commercial system (Interacoustic Eclipse TM) device during passive listening to a 60dB auditory stimulus and active speaking conditions
Difference in amplitude of cortical auditory evoked potentials in children with stuttering compared to children who do do not stutter | baseline: before intervention
  Measuring amplitude in microvolt of P1, N1 using the commercial system (Interacoustic Eclipse TM)
Change in amplitude of cortical auditory evoked potentials in children with stuttering due to stuttering intervention program | immediately after intervention
  Measuring amplitude in microvolt of P1, N1 in the group who stutter after intervention using the commercial system (Interacoustic Eclipse TM) device during passive listening to a 60dB auditory stimulus and active speaking conditions

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Abdou Mustafa, PhD, Study Chair — Otorhinolaryngology department,Faculty of Medicine, Alexandria University; Mohamed A Talaat, PhD, Study Chair — Otorhinolaryngology department,Faculty of Medicine, Alexandria University; Engy S Elhakeem, PhD, Study Director — Otorhinolaryngology department,Faculty of Medicine, Alexandria University; Alaa M Radwan, MS, Principal Investigator — Otorhinolaryngology department, Faculty of Medicine, Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria universtiy, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there would be a plane to make IPD available
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: anticipated 4 to 6 months for the data to be available
Access Criteria: Through the Email Address A_abdelhamed14@alexmed.edu.eg

REFERENCES:
- [Background] Ismail N, Sallam Y, Behery R, Al Boghdady A. Cortical auditory evoked potentials in children who stutter. Int J Pediatr Otorhinolaryngol. 2017 Jun;97:93-101. doi: 10.1016/j.ijporl.2017.03.030. Epub 2017 Apr 3. PMID 28483259
- [Background] Abdou R. Assessment of Egyptian children who stutter using the standardized Arabic form of the Test of Childhood Stuttering. The Egyptian Journal of Otolaryngology. 2015;31(3):180-7.
- [Background] Duncan CC, Barry RJ, Connolly JF, Fischer C, Michie PT, Naatanen R, Polich J, Reinvang I, Van Petten C. Event-related potentials in clinical research: guidelines for eliciting, recording, and quantifying mismatch negativity, P300, and N400. Clin Neurophysiol. 2009 Nov;120(11):1883-1908. doi: 10.1016/j.clinph.2009.07.045. Epub 2009 Sep 30. PMID 19796989
- [Result] Packman A, Attanasio J, editors. A model of the mechanisms underpinning early interventions for stuttering. Seminar presentation at the annual convention of the American Speech-Language and Hearing Association Philadelphia, USA; 2010.
- [Result] Cone-Wesson B, Wunderlich J. Auditory evoked potentials from the cortex: audiology applications. Curr Opin Otolaryngol Head Neck Surg. 2003 Oct;11(5):372-7. doi: 10.1097/00020840-200310000-00011. PMID 14502069